CLINICAL TRIAL: NCT07192198
Title: Efficacy of Inhaled Methoxyflurane (Penthrox) as Adjunct for Urologic Procedures Under Local Anesthetic: A Pilot Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Premal Patel, MD, Assistant Professor, Department of Surgery. Director, Undergraduate Urologic Medical Education, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS26348
Record Dates: First submitted 2024-02-16; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Scrotum Disease; Hydrocele Male; Spermatocele; Scrotal Hematocele; Anesthesia, Local
MeSH Terms: conditions — Spermatocele; Hematocele | interventions — Methoxyflurane

STUDY DESIGN:
Intervention Model Description: Double blinded, placebo controlled, randomized trial. Two arms, one is the intervention arm which will receive Penthrox and local anesthesia infiltration while the control arm will receive local anesthesia infiltration.
Who Masked: Participant, Care Provider
Masking Description: The surgeon and patient are both blinded to which cream is being utilized, whether it be Penthrox, or a control. Investigators and study personnel are not blinded to this.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention arm-Penthrox (Experimental): Participants can begin using penthrox 10 minutes prior to procedure start, given its median onset time of 5 minutes
  Interventions: Drug: Methoxyflurane
- Control arm (Placebo Comparator): Patients in the control arm will only receive local infiltration.
  Interventions: Other: Control

INTERVENTIONS:
Drug: Methoxyflurane — Penthrox is a brand name for a drug called methoxyflurane. It is an inhaled analgesic (pain-relieving) agent used primarily for the relief of moderate to severe pain, typically in emergency medical situations or during minor medical procedures. Penthrox is administered by inhaling the vapors through a hand-held inhaler device. It acts quickly to provide pain relief and has a relatively short duration of action.
  Arms: Intervention arm-Penthrox
Other: Control — This intervention will be the control group, only receiving local infiltration.
  Arms: Control arm

SUMMARY:
We wish to perform a prospective randomized controlled pilot study at the Men's Health Clinic and Health Science's Centre to assess whether or not the use of Penthrox as an adjunct to LA is associated with improved pain tolerance and anxiety levels than local anesthetic alone

DETAILED DESCRIPTION:
This non-blinded, randomized controlled trial is to be conducted at both the Men's Health Clinic and Health Sciences Centre in Winnipeg, Manitoba. All eligible patients between the ages of 18-65, undergoing andrology and male infertility under local anesthetic or select endourology procedures under loco-sedation, will be invited to participate in the study. Patients will be excluded if; history of substance use disorder, history renal impairment, history of liver dysfunction, previous hypersensitivity to Penthrox or related agents, personal or family history of malignant hypothermia. They will be randomly assigned in a 1:1 ratio using a computer-generated random list. For penoscrotal cases, patient will be randomized to Penthrox + local infiltration of 50/50 lidocaine and bupivacaine mixture vs local infiltration alone. For select endourology procedures, patients will be randomized to Penthrox + topical local anesthetic vs IV sedation + topical anesthetic. Participants may begin using the Penthrox 10 minutes prior to procedure start given its median time of onset of 5 minutes. In the post-operative recovery area, patient will be asked to complete a questionnaire related to pain and anxiety of procedure.

Baseline characteristics such as age, use of analgesics, prior history of procedure under loco-sedation, history of chronic pain, baseline pain level (Brief Pain Inventory), pre-procedural anxiety (State Trait Anxiety Inventory) will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing hydrocelectomy, spermatocelectomy, epididymectomy, testicular biopsy, scrotal lesion or cyst excision under local anesthesia alone will be included.

Exclusion Criteria:

* Patients will be excluded if their procedure was to be performed with sedatives (e.g., inhaled nitrous oxide gas, oral, or IV sedation) or did not provide consent to be randomized

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-04-17 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
Pain with local anesthetic infiltration | Immediately post-infiltration, intraoperatively
  Using a visual analogue pain scale [range 0-10; 0 = no pain, 10 = maximal pain], pain will be assessed as reported by the patient when the local anesthetic injection is administered
Procedural pain | Immediately post-operation
  Using a visual analogue pain scale [range 0-10; 0 = no pain, 10 = maximal pain], pain will be assessed as reported by the patient post-operatively to determine their pain

CONTACTS AND LOCATIONS:
Locations (1):
- Men's Health Clinic, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No